CLINICAL TRIAL: NCT06262997
Title: Effectiveness of Pilates and Kinesiotape Applications in Office Workers With Neck Pain
Brief Title: Effectiveness of Pilates and Taping in Office Workers With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Ali MUTLU, Research Assistant of Department of Physiotherapy and Rehabilitation, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TU-FTR-AMUTLU-2
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-02

CONDITIONS: Neck Pain
Keywords: Neck Pain; Office Workers; Postural Awareness; Quality of Daily Life; Range of Motion
MeSH Terms: conditions — Neck Pain | interventions — Exercise Movement Techniques; Athletic Tape

STUDY DESIGN:
Intervention Model Description: One group will receive only pilates training. Other group participants will receive kinesiobant application in addition to pilates training.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor who will administer the pretest and post-test is blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates (Active Comparator): Participants will receive an average of 1 hour of pilates training accompanied by a physiotherapist for 8 weeks, 2 days a week in groups of 2-3 people.
  Interventions: Other: Pilates
- Pilates and Kinesiotape (Experimental): They will receive exactly the same Pilates training as the patients in the Pilates group and in addition kinesio tape will be applied.
  Interventions: Other: Pilates and Kinesiotape

INTERVENTIONS:
Other: Pilates — Pilates training will be given to groups of 3 people for 8 weeks, 2 days a week. Exercises will start with 10-12 repetitions and the number of repetitions will be increased to 20 starting from the 4th week. Before the Pilates training, basic principles such as breathing, concentration, focusing on the center, control, precision and fluid movement will be taught in a special session to inform individuals about the training principles and exercises. Each exercise will be demonstrated by the physiotherapist and cues such as tactile, verbal and imagery will be used to control the participants throughout the training. The difficulty level of Pilates training will be progressed by changing body positions, exercise ball and band use according to the performance of the patients and Pilates principles. The exercise program will start with warm-up exercises and end with 40 minutes of basic Pilates exercises followed by cooling exercises.
  Arms: Pilates
Other: Pilates and Kinesiotape — Patients in the Pilates and Kinesiotape group will receive exactly the same Pilates training as in the Pilates group. At the end of each exercise session, Kinesio Tex Gold FP elastic tape (5 cm) will be applied with mechanical correction technique for postural correction and the tape will be renewed in each session. Waterproof, porous, adhesive, 0.5 mm thick tape will be applied to the upper trapezius.
  Arms: Pilates and Kinesiotape

SUMMARY:
The aim of this study is to investigate the effectiveness of pilates and kinesiotape applications in office workers with neck pain. In this direction, neck pain and disability, pain threshold, muscle strength, range of motion, core endurance, postural awareness and quality of life will be evaluated.

DETAILED DESCRIPTION:
The aim of this randomized controlled experimental study was to investigate the effectiveness of Pilates and kinesiotape in office workers with neck pain. In this study where a total of 42 office workers will be followed for 8 weeks, individuals will be randomly divided into two groups. The training groups will consist of 3 people each. The control group will receive only Pilates training and the experimental group will receive kinesio taping in addition to Pilates training. Individuals will be analyzed for neck pain and disability, pain threshold, muscle strength, range of motion, core endurance, postural awareness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have been office workers for at least 1 year
* Using a computer at a desk for at least 3 hours a day
* Having neck pain for more than 6 weeks
* Having neck pain rated at or above 3/10 on a visual analog scale

Exclusion Criteria:

* Having neurological and rheumatologic chronic diseases
* Having received physical therapy in the last 6 months
* Having a history of trauma to the spine
* Having a history of surgery in the cervical spine
* Having diagnosed cervical/lumbar disc and spine pathologies
* Having an allergic reaction to taping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 2 months
  It will be used to assess neck disability. The scale is used to show the effects of neck pain on the daily lives of individuals. The Turkish validity and reliability scale consists of 10 sections including pain intensity, self-care, lifting, reading, headache, concentration, work life, driving, sleep and leisure time activities. Each section is scored between 0 (no disability) and 5 (full disability). Scores from the scale range between 0-50 and the higher the score, the higher the level of disability. According to the scale, a score of 0-4 is considered as no disability, 5-14 as mild disability, 15-24 as moderate disability, 25-34 as severe disability and 35 and above as complete disability.

SECONDARY OUTCOMES:
Pain PressureThreshold | 2 months
  Pressure pain threshold refers to the lowest force that must be applied for pressure sensation to be transformed into pain sensation. A pressure algometer will be used to measure the pressure pain threshold. The pain threshold will be measured from the upper part of the trapezius muscle and the tibialis anterior muscle trunk
Muscle Strength | 2 months
  Assessment of muscle strength is an important clinical assessment for patients with neurological, muscular and/or skeletal diseases. Such clinical information provides a basis of knowledge when the patient first presents. If a treatment plan is subsequently followed, muscle strength assessments can help determine treatment efficacy. In this study, neck muscle strength will be assessed with a mechanical push pull dynamometer.
Range of Motion | 2 months
  Neck (cervical region) joint motion consists of flexion, extension, lateral flexion and rotation. The use of specific tools to assess range of motion (ROM) allows for an objective and standardized assessment during follow-up. Inclinometer is one of the commonly used measurement tools for neck ROM measurements. A inclinometer will be used to assess neck flexion and lateral flexion, and neck rotation.
Prone Bridge Test | 2 months
  Static endurance of the "core" muscles will be evaluated with the "prone bridge" test. In the prone bridge test, individuals are asked to lift their torso upwards by placing their weight on their forearms and toes in the prone, elbows flexed position. Measurements are recorded in seconds using a stopwatch, and the test is terminated when the test position is broken. Each measurement will be performed 2 times and the best measurement will be used for statistical analysis.
Sits Up Test: | 2 months
  The assessment of the dynamic endurance of the "core" muscles will be performed with the Sits-up test. The number of times the individuals can perform each test for 30 seconds will be recorded. In the sit-up test, individuals are asked to perform trunk flexion with knees in flexion position and feet stabilized.
Postural Habits and Awareness Scale | 2 months
  It was developed by Bayar et al. to assess the postural habits and awareness of individuals. The scale is a 5-point Likert scale and consists of a total of 19 items, 7 items evaluating postural habits and 12 items evaluating postural awareness. The score that can be obtained from the scale is in the range of 0-95 and a high score indicates a good posture and awareness.
Short Form 36 | 2 months
  It is one of the scales frequently used to measure quality of life. The scale consists of 8 subscales (physical function, social function, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain and general perception of health) and 36 items in total.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Göz, Study Director — Tarsus University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No